CLINICAL TRIAL: NCT01884974
Title: A Case Control Study of the Prevalence of Pulmonary Hypertension in Patients With Myeloproliferative Diseases, and Correlation Between Patients Epidemiologic and Clinical Status and the Development of Pulmonary Hypertension.
Brief Title: A Case Control Study of the Prevalence of Pulmonary Hypertension in Patients With Myeloproliferative Diseases.
Acronym: PH-MPD1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Shoshan Perek, Dr Shoshan Perek, Carmel Medical Center
Other Study IDs: CMC-12-0060-CTIL
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Myeloproliferative Disease; Pulmonary Hypertension
Keywords: Myeloproliferative disease; Pulmonary Hypertension
MeSH Terms: conditions — Myeloproliferative Disorders; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- myeloproliferative disease: Patients with Myeloproliferative Diseases as specified under inclusion and exclusion criteria
  Interventions: Other: myeloproliferative disease

INTERVENTIONS:
Other: myeloproliferative disease — Echocardiogram, demographic data, St George respiratory questioner

SUMMARY:
Pulmonary hypertension (PH) is defined as a group of diseases characterised by an elevated mean pulmonary artery pressure (Ppa) ≥25 mmHg at rest. Recently, chronic myeloproliferative diseases (CMPD) associated with pulmonary hypertension were included in the group 5 category, corresponding to PH for which the aetiology is unclear and/or multifactorial. CMPD include chronic myelogenous leukaemia, chronic neutrophilic leukaemia and chronic eosinophilic leukaemia (which primarily express a myeloid phenotype and polycythaemia vera), idiopathic myelofibrosis, and essential thrombocytosis in which erythroid or megakaryocytic hyperplasia predominates.

The purpose of this research:

1. Assess Prevalence of PH in patients with CMPD in Northern Israel
2. Describe the demographics and clinical course in patients with CMPD who are diagnosed with PH.

DETAILED DESCRIPTION:
study will include the following:

* sex
* age
* BMI
* ethnicity
* age diagnosed with Myeloproliferative disease
* clinical manifestations of the myeloproliferative disease
* JAK2 mutation
* known hematological complications

ELIGIBILITY:
Inclusion Criteria:

1) consenting patients diagnosed with a myeloproliferative disease

Exclusion Criteria:

1) Refusal to have an echocardiogram or answer the St. George respiratory questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with Myeloproliferative disease and followed up at the Carmel Hematology Unit
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
pulmonary hypertension | 1 year
  all patients with myeloproliferative diseases in the study will be evaluated by an echocardiogram. Pulmonary hypertension will be considered when the average pulmonary arterial pressure is equal or above 25 mmHg.

SECONDARY OUTCOMES:
St George Respiratory Questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shoshan Perek, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Pulmonology Institute, Carmel Medical Center, Haifa, Israel